CLINICAL TRIAL: NCT03065127
Title: Investigating Therapies for Freezing of Gait Targeting the Cognitive, Limbic, and Sensorimotor Domains
Brief Title: Investigating Therapies for Freezing of Gait
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Life Financial Movement Disorders Research and Rehabilitation Centre (Other)
Responsible Party: Principal Investigator, Rebecca Chow, Primary Investigator, Sun Life Financial Movement Disorders Research and Rehabilitation Centre
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SunLife
Record Dates: First submitted 2017-02-09; First posted 2017-02-27 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Parkinson Disease; Gait Disorders, Neurologic
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic | interventions — Cognitive Training; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Training (Experimental): Participants will independently complete cognitive exercises on the "Smartbrain Pro" computer software. These exercises aim to train different aspects of executive function. The difficulty level of each exercise will increase relative to each participant's progress. Sessions will last for one hour, occurring twice weekly for a period of 4 weeks.
  Interventions: Behavioral: Cognitive Training
- Cognitive Behavioural Therapy (Experimental): Participants will undergo one-on-one sessions of cognitive-behavioural therapy (CBT) working with a therapist to establish an individualized CBT plan which will focus on symptoms of anxiety. Participants will complete a total of eight one-hour sessions over 4 weeks.
  Interventions: Behavioral: Cognitive Behavioural Therapy
- Proprioceptive Training (Experimental): Participants will complete one-on-one sessions a target matching proprioceptive training protocol using their upper and lower limbs. For the upper limb target-reaching task, participants will be seated in front of a surface marked with ten targets. They will first visualize a specified target, then blindfolded and asked to reach towards that target with the blindfold on. The blindfold will then be removed allowing participants to view their performance relative to the target. This task will be repeated for the remaining targets on both sides and for both upper and lower limbs. Participants will complete a total of eight one-hour sessions over 4 weeks.
  Interventions: Behavioral: Proprioceptive Training

INTERVENTIONS:
Behavioral: Cognitive Training — Training the cognitive domain may be accomplished by training various cognitive and executive functions with guided practice focusing on specific skills (e.g. visuospatial processing, executive function, memory, language, and attention). Cognitive training has been demonstrated to be efficacious in several studies in individuals with PD. Given the potential cognitive contribution to FOG episodes, this type of therapy may alleviate FOG by potentially improving upon planning, set-shifting, and/or response inhibition.
  Arms: Cognitive Training
Behavioral: Cognitive Behavioural Therapy — CBT has been demonstrated to be effective in the remediation of anxiety in individuals with PD. This may be beneficial to individuals experiencing FOG, given the evidence that anxiety may provoke FOG. During periods of elevated anxiety (e.g. walking in a threatening environment), freezers will be able to more efficiently process this limbic load resulting in greater resources available for movement control.
  Arms: Cognitive Behavioural Therapy
Behavioral: Proprioceptive Training — Currently, studies investigating proprioceptive training as a treatment in PD are limited. However, this type of training has potential by improving proprioceptive processing. It would be expected that due to this training, when sensorimotor processing is challenged during locomotion (e.g. by removing visual feedback and preventing compensation of proprioception deficits), freezers would experience less decrements to gait due to an enhanced ability to process sensorimotor demands.
  Arms: Proprioceptive Training

SUMMARY:
Freezing of gait (FOG) is arguably one of the most debilitating motor symptoms experienced by individuals with Parkinson's disease (PD). FOG may be caused by an overload of cognitive, limbic, and sensorimotor system activity in the basal ganglia. Therefore, the purpose of this study is to evaluate cognitive, limbic, and sensorimotor therapies in individuals with FOG. Participants in this study will undergo all three types of treatments in a randomized counterbalanced order. Each treatment will occur in 1 hour sessions, twice weekly for a period of 4 weeks.

DETAILED DESCRIPTION:
Freezing of gait (FOG) is arguably one of the most debilitating motor symptoms experienced by individuals with Parkinson's disease (PD), and negatively impacts quality of life (Walton et al., 2015). Furthermore, advanced FOG does not respond well to treatments commonly used in Parkinson's disease (Nutt et al., 2011), therefore warranting the use of adjunct treatment options. The development of potential treatment strategies for FOG should focus on the underlying mechanism. The cross-talk model of FOG proposes that FOG may be caused by an overload of cognitive, limbic, and sensorimotor system activity in the basal ganglia, resulting in a depletion of dopaminergic resources, leading to FOG (Lewis & Barker, 2009). Hence, based on the cross-talk model, treatments targeting the cognitive, sensorimotor and limbic systems independently may lead to a reduction in FOG episodes. Previous studies have demonstrated the efficacy of therapies targeting these domains in PD and healthy individuals, however, these have yet to be explored in FOG. Therefore, the purpose of this study is to evaluate cognitive, sensorimotor, and limbic therapies in individuals with FOG.

This study will employ a within-subjects design, in which participants will undergo all three treatments in a randomized counterbalanced order. Sessions for each type of treatment will occur for 1 hour, twice weekly for a period of 4 weeks. Participants will also undergo pre- and post-test assessments prior to and following each 4-week treatment period. The cognitive training will utilize the "Smartbrain Pro" computer software, which has previously demonstrated efficacy in individuals with Parkinson's disease (Paris et al., 2011). The sensorimotor training group will participate in proprioceptive training of the upper and lower limbs. This training will entail a target matching task, in which participants will produce active and self-defined movements while blindfolded (i.e. without visual feedback). The limbic training group will undergo cognitive behavioural therapy (CBT) focusing solely on anxiety symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Either gender
* Diagnosed with idiopathic PD by a Neurologist
* Self-reported FOG with the use of UPDRS-II (Question 14)
* Confirmation of present FOG by a movement disorder specialist
* Able to walk 10 meters, unassisted
* Able to understand English instructions

Exclusion Criteria:

* A neurological disease other than PD
* Peripheral neuropathy
* Clinically diagnosed with dementia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Gait Assessment | Change from Baseline at 4 weeks of first treatment phase
  Participants will walk approximately 9.75 metres for 12 trials. Recording of kinematic data will be done with eight Optotrak® cameras (Northern Digital, NDI, Waterloo, Ontario). Spatiotemporal gait parameters will be analyzed from this assessment.
Gait Assessment | Change from Baseline at 4 weeks of second treatment phase
  Participants will walk approximately 9.75 metres for 12 trials. Recording of kinematic data will be done with eight Optotrak® cameras (Northern Digital, NDI, Waterloo, Ontario). Spatiotemporal gait parameters will be analyzed from this assessment.
Gait Assessment | Change from Baseline at 4 weeks of third treatment phase
  Participants will walk approximately 9.75 metres for 12 trials. Recording of kinematic data will be done with eight Optotrak® cameras (Northern Digital, NDI, Waterloo, Ontario). Spatiotemporal gait parameters will be analyzed from this assessment.

SECONDARY OUTCOMES:
Stroop Test | Pre-intervention and Post-intervention at week 4 of first treatment phase
  This test assesses inhibitory control and will be administered in a paper-based format.
Trail-making test | Pre-intervention and Post-intervention at week 4 of first treatment phase
  This will also be administered in a paper-based format. This test will assess visuospatial function and set-shifting ability.
Stroop Test | Pre-intervention and Post-intervention at week 4 of second treatment phase
  This test assesses inhibitory control and will be administered in a paper-based format.
Trail-making test | Pre-intervention and Post-intervention at week 4 of second treatment phase
  This will also be administered in a paper-based format. This test will assess visuospatial function and set-shifting ability.
Stroop Test | Pre-intervention and Post-intervention at week 4 of third treatment phase
  This test assesses inhibitory control and will be administered in a paper-based format.
Trail-making test | Pre-intervention and Post-intervention at week 4 of third treatment phase
  This will also be administered in a paper-based format. This test will assess visuospatial function and set-shifting ability.
Passive Joint Angle Matching | Pre-intervention and Post-intervention at week 4 of first treatment phase
  This task will be assessed in order to evaluate proprioceptive functioning.
Passive Joint Angle Matching | Pre-intervention and Post-intervention at week 4 of second treatment phase
  This task will be assessed in order to evaluate proprioceptive functioning.
Passive Joint Angle Matching | Pre-intervention and Post-intervention at week 4 of third treatment phase
  This task will be assessed in order to evaluate proprioceptive functioning.
Parkinson Anxiety Scale | Pre-intervention and Post-intervention at week 4 of first treatment phase
  The Parkinson Anxiety Scale (PAS), which is a self-report questionnaire used to assess anxiety levels, will be administered to participants. This tool has demonstrated good concurrent validity in individuals with PD against other existing anxiety scales (Leentjens et al., 2014).
Parkinson Anxiety Scale | Pre-intervention and Post-intervention at week 4 of second treatment phase
  The Parkinson Anxiety Scale (PAS), which is a self-report questionnaire used to assess anxiety levels, will be administered to participants. This tool has demonstrated good concurrent validity in individuals with PD against other existing anxiety scales (Leentjens et al., 2014).
Parkinson Anxiety Scale | Pre-intervention and Post-intervention at week 4 of third treatment phase
  The Parkinson Anxiety Scale (PAS), which is a self-report questionnaire used to assess anxiety levels, will be administered to participants. This tool has demonstrated good concurrent validity in individuals with PD against other existing anxiety scales (Leentjens et al., 2014).
Unified Parkinson's disease Rating Scale Motor Subsection (UPDRS-III) | Pre-intervention and Post-intervention at week 4 of first treatment phase
  A clinician administered assessment which evaluates individuals' motor symptom severity
Unified Parkinson's disease Rating Scale Motor Subsection (UPDRS-III) | Pre-intervention and Post-intervention at week 4 of second treatment phase
  A clinician administered assessment which evaluates individuals' motor symptom severity
Unified Parkinson's disease Rating Scale Motor Subsection (UPDRS-III) | Pre-intervention and Post-intervention at week 4 of third treatment phase
  A clinician administered assessment which evaluates individuals' motor symptom severity
New Freezing of Gait Questionnaire (NFOGQ) | Pre-intervention and Post-intervention at week 4 of first treatment phase
  Participants will be asked to complete the New Freezing of Gait Questionnaire (NFOGQ) questionnaire developed by Nieuwboer and colleagues (2009). This provides a self-reported measure of frequency and duration of FOG episodes. This tool has been validated and proven to be highly reliable in individuals with PD, as well as assessing treatment interventions for FOG.
New Freezing of Gait Questionnaire (NFOGQ) | Pre-intervention and Post-intervention at week 4 of second treatment phase
  Participants will be asked to complete the New Freezing of Gait Questionnaire (NFOGQ) questionnaire developed by Nieuwboer and colleagues (2009). This provides a self-reported measure of frequency and duration of FOG episodes. This tool has been validated and proven to be highly reliable in individuals with PD, as well as assessing treatment interventions for FOG.
New Freezing of Gait Questionnaire (NFOGQ) | Pre-intervention and Post-intervention at week 4 of third treatment phase
  Participants will be asked to complete the New Freezing of Gait Questionnaire (NFOGQ) questionnaire developed by Nieuwboer and colleagues (2009). This provides a self-reported measure of frequency and duration of FOG episodes. This tool has been validated and proven to be highly reliable in individuals with PD, as well as assessing treatment interventions for FOG.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Chow, BSc, Principal Investigator — Sun Life Financial Movement Disorders Research and Rehabilitation Centre
Locations (1):
- Sun Life Financial Movement Disorders Research and Rehabilitation Centre, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chow R, Tripp BP, Rzondzinski D, Almeida QJ. Investigating Therapies for Freezing of Gait Targeting the Cognitive, Limbic, and Sensorimotor Domains. Neurorehabil Neural Repair. 2021 Mar;35(3):290-299. doi: 10.1177/1545968321992331. Epub 2021 Feb 9. PMID 33559531